CLINICAL TRIAL: NCT05475327
Title: Effects of Progressive Relaxation Exercises on Low Back Pain and Insomnia in the Third Trimester of Pregnancy
Brief Title: Relaxation Exercises for Low Back Pain and Insomnia in the Third Trimester of Pregnancy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REC/RCR & AHS/22/0512
Record Dates: First submitted 2022-07-24; First posted 2022-07-26 (Actual); Last update posted 2023-09-18 (Actual); Status verified 2023-09

CONDITIONS: Low Back Pain
Keywords: Pregnancy; Respiratory training; Sleep disturbance
MeSH Terms: conditions — Low Back Pain; Parasomnias

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional Physical Therapy (Other): Heat therapy and education regarding back care management.
  Interventions: Other: Conventional Physical Therapy
- Relaxation exercises (Experimental): Progressive relaxation exercises along with Deep Breathing exercises.
  Interventions: Other: Relaxation exercises

INTERVENTIONS:
Other: Conventional Physical Therapy — Heating pad
  A total of 3 sessions per week were given for 15 to 20 mins
  Arms: Conventional Physical Therapy
Other: Relaxation exercises — The experimental group was given Progressive relaxation exercises along with Deep breathing exercises.
  A total of 3 sessions per week were given for 15 to 20 mins.
  Arms: Relaxation exercises

SUMMARY:
The role of progressive muscle exercises has been widely explored. However, limited studies report its effectiveness in pregnant women in their third trimester suffering from pain and insomnia that may or may not be due to that pain. This study aims to determine the effects of relaxation exercises on low back pain and insomnia.

DETAILED DESCRIPTION:
In 2021 the research says that most women experience pubic pain, hip pain, knee pain, leg cramps, carpal tunnel syndrome, De Quervain's tenosynovitis, or at least one of these symptoms during pregnancy and approximately one-quarter of them have a temporary disability. Symptoms of LBP could start from early in pregnancy until giving birth, but usually, the pain becomes more severe during the third semester of pregnancy and is described as a dull pain. In most cases of LBP, the pain does not radiate to other parts of the body. The exercise was found to be a very common practice used to decrease LBP and the majority of the relative studies were categorized as of high methodological quality. The exercise components of the interventions included strength and stretching, endurance training, pelvic tilt exercises, stretching and mild isometric abdominal contractions, progressive muscle relaxation exercises accompanied by music as well as aerobic and stretching exercises.

Another research in 2021 describe that one of the most common complaints during pregnancy is sleep disorders, such as insomnia, frequently waking up at night, high drowsiness during the day, mood swings, and unusual feelings during sleep results of the present study showed that counseling with a spiritual approach was effective in improving the sleep quality in pregnant women. In the intervention group, the mean score of sleep quality decreased in the second and third trimesters compared to the control group. In the present study, spiritual content counseling had a significant effect on all areas of sleep quality, except for habitual sleep efficiency.

In 2018 one of research says that physiological and psychological changes in the third trimester of pregnancy make falling asleep at night more difficult for pregnant women. Studies also show that relaxation exercises reduce psychological tension, stress, and pain. The pregnant women in the relaxation exercises group of the present study reported falling asleep more comfortably as a result of the decrease in muscle tension, stress, and pain perception. The four-week relaxation exercises improved subjective sleep latency, duration, habitual sleep efficiency, sleep disturbances, daytime dysfunction, and sleep quality of the pregnant women in the third trimester.

Another research in 2018 on the effects of breathing exercises on insomnia. This study finding revealed that, pre-intervention more than half of the pregnant women experienced severe insomnia this may be attributed to the inflammation process of pregnancy and the effect of pregnancy physiological and psychological changes and discomforts on the sleep cycle. The present study revealed that the total score of insomnia decreased for the majority of pregnant women after practicing walking with deep breathing exercises. This can be attributed to the positive effect of exercises i.e walking or breathing exercises on the overall health either physical or psychological by improving physical fitness, increasing the blood supply and the circulation to the brain to enhance the sleep cycle, and improving the quality of sleep and decrease the insomnia symptoms. It has a positive effect on the severity of insomnia during the third trimester of pregnancy, tension, and fatigue relief.

Another research in 2014 says that relaxation therapy and progressive muscle relaxation (PMR) are forms of complementary and alternative medicine often used in pregnancy. There are several reasons why this therapy might produce the observed benefit. PMR-induced reduction in anxiety and decreased perception of pain may eventually improve QOL status in pregnant women. In one study, PMR intervention was compared with massage in pregnant women with leg and back pain. In that study, leg pain decreased significantly after the first and last treatments in both the PMR and massage groups, but back pain decreased only in the massage group. Pain decreased over time during the study in the intervention group, whereas the pain scores (and perceived pain) in the control group increased gradually. LBP is one of the most common symptoms in pregnancy. We conclude that PMR training can reduce LBP and improve QOL in pregnant women.

Most of the research was conducted on low back pain with pelvic girdle pain, the effect of relaxation exercises with music on low back pain, the effect of relaxation exercises on insomnia, and quality of life. The objective of this research is to determine the effect of progressive relaxation exercises on low back pain and insomnia in the third trimester of pregnancy and show the combined effect of relaxation. Reviewing the previous literature on the effects of exercises on low back pain and insomnia provides sufficient data but there is not enough data on the effects of a combination of both exercise on insomnia and low back pain.

ELIGIBILITY:
Inclusion Criteria:

* Uncomplicated pregnancies
* Chronic back pain for at least 3 months without radiation to legs

Exclusion Criteria:

* High-risk pregnancy
* Previous spinal surgery
* Structural spinal deformities like scoliosis or Spondylolisthesis
* Diagnosed depression or anxiety
* Diagnosed Disk herniation
* Rheumatic conditions involving the spine

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 30 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2022-08-01 (Actual); Study Completion 2022-08-01 (Actual)

PRIMARY OUTCOMES:
Roland-Morris Low Back Pain and Disability Questionnaire | 6th week
  Changes from baseline the Roland-Morris Questionnaire (RMQ) is a self-administered disability measure in which greater levels of disability are reflected by higher numbers on a 24-point scale. The RMQ has been shown to yield reliable measurements, which are valid for inferring the level of disability and to be sensitive to change over time for groups of patients with low back pain.
  Roland and Morris did not provide descriptions of the varying degrees of disability (eg, 40%-60% is a severe disability). A clinical improvement over time can be graded based on the analysis of serial questionnaire scores. If, for example, at the beginning of treatment, a patient's score was 12 and, after treatment, their score was 2 (10 points of improvement), we would calculate an 83% (10/12 x 100) improvement.

SECONDARY OUTCOMES:
Numeric Pain Rating Scale (NPRS) | 6th week
  Changes from baseline the Numeric Pain Rating Scale (NPRS) is a unidimensional measure of pain intensity in adults. The 11-point numeric scale ranges from '0' representing one pain extreme (e.g. "no pain") to '10' representing the other pain extreme (e.g. "pain as bad as you can imagine" or "worst pain imaginable")
Insomnia Severity Index | 6th week
  Changes from baseline the Insomnia Severity Index has seven questions. The seven answers are added up to get a total score.
  Total score categories:
  0-7 = No clinically significant insomnia 8-14 = Subthreshold insomnia 15-21 = Clinical insomnia (moderate severity) 22-28 = Clinical insomnia (severe)

CONTACTS AND LOCATIONS:
Overall Officials: Afifa Safdar, PhD*, Principal Investigator — Riphah International University
Locations (1):
- Bashir Hospital, Sialkot, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Akmese ZB, Oran NT. Effects of Progressive Muscle Relaxation Exercises Accompanied by Music on Low Back Pain and Quality of Life During Pregnancy. J Midwifery Womens Health. 2014 Sep-Oct;59(5):503-9. doi: 10.1111/jmwh.12176. Epub 2014 Jun 25. PMID 24965313
- [Background] Sadeghi B, Sirati-Nir M, Hajimini Z, Ebadi A, Ali-Asgari M. Comparing the Effects of Progressive Muscle Relaxation and Physical Activity on Pregnant Women's General Health. Iran J Nurs Midwifery Res. 2018 Jul-Aug;23(4):298-304. doi: 10.4103/ijnmr.IJNMR_54_17. PMID 30034491
- [Background] Ozkan SA, Rathfisch G. The effect of relaxation exercises on sleep quality in pregnant women in the third trimester: A randomized controlled trial. Complement Ther Clin Pract. 2018 Aug;32:79-84. doi: 10.1016/j.ctcp.2018.05.008. Epub 2018 May 26. PMID 30057064
- [Background] Koukoulithras I Sr, Stamouli A, Kolokotsios S, Plexousakis M Sr, Mavrogiannopoulou C. The Effectiveness of Non-Pharmaceutical Interventions Upon Pregnancy-Related Low Back Pain: A Systematic Review and Meta-Analysis. Cureus. 2021 Jan 30;13(1):e13011. doi: 10.7759/cureus.13011. PMID 33728108
- [Background] Childs JD, Piva SR, Fritz JM. Responsiveness of the numeric pain rating scale in patients with low back pain. Spine (Phila Pa 1976). 2005 Jun 1;30(11):1331-4. doi: 10.1097/01.brs.0000164099.92112.29. PMID 15928561
- [Background] Bastien CH, Vallieres A, Morin CM. Validation of the Insomnia Severity Index as an outcome measure for insomnia research. Sleep Med. 2001 Jul;2(4):297-307. doi: 10.1016/s1389-9457(00)00065-4. PMID 11438246
- [Background] Roland M, Fairbank J. The Roland-Morris Disability Questionnaire and the Oswestry Disability Questionnaire. Spine (Phila Pa 1976). 2000 Dec 15;25(24):3115-24. doi: 10.1097/00007632-200012150-00006. No abstract available. PMID 11124727